CLINICAL TRIAL: NCT01742975
Title: A Randomized Study Evaluating the Efficacy of the Synthetic Adhesive Solution Ifabond, in Reducing Seroma Formation Post Surgery in Breast Cancer Patients, When Used in Partial Mastectomy With or Without Axillary Lymph Node Dissection
Brief Title: Efficacy Study of Ifabond in Breast Cancer Surgery
Acronym: Ifabond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-15 ONC HAP
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2016-08

CONDITIONS: Breast Cancer; Lymphocele
MeSH Terms: conditions — Breast Neoplasms; Lymphocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Applying Ifabond (Experimental): The synthetic adhesive solution Ifabond, will be applied at the end of conventional breast cancer surgery for arm A patients.
  Interventions: Device: IFABOND (TM)
- Arm B: without Ifabond (No Intervention): The synthetic adhesive solution Ifabond, will not be applied at the end of conventional breast cancer surgery in arm B patients.

INTERVENTIONS:
Device: IFABOND (TM) — The synthetic adhesive solution Ifabond, will be applied at the end of conventional breast cancer surgery for arm A patients
  Other Names: An authorized device with CE labeling.
  Arms: Arm A: Applying Ifabond

SUMMARY:
A randomized prospective simple-blind interventional study evaluating the efficacy of the synthetic adhesive solution "Ifabond", in patients undergoing breast cancer surgery. The main objective of this study is to determine if the application of Ifabond, in addition to the conventional method of breast surgery, reduces the postoperative seroma formation. The secondary objective is to assess quality of life immediately after surgery, and the need for needle aspiration of the axilla, when using Ifabond.

DETAILED DESCRIPTION:
Breast cancer patients will be selected at their preoperative visit with the surgeon, who will inform them about the study and answer their questions.

Patients who consent to participate will be randomized to one of two arms:

1. Arm A: Applying Ifabond
2. Arm B: Without Ifabond

Patients will be stratified according to these two criteria:

1. Axillary Lymph Node Dissection planned (ALND)
2. Body Mass Index (BMI)

The following parameters will be measured:

* ECOG status and Blood Pressure at day 3(day 7 in case of ALND), day 15 and day 30 post surgery
* Volume of drainage at day 3 and at (day 7 in case of ALND)post surgery
* Discomfort alleged by the patient at day 3(day 7 in case of ALND), day 15 and day 30 post surgery
* Lymphocele volume measured by ultrasound at day 15 and day 30 post surgery
* If the volume is ≥ 100cc, a needle aspiration will be performed, and the volume of aspirate will be documented.
* Adverse events and concomitant medications will be collected throughout the study until 30 days after the last ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* "Eastern Cooperative Oncology Group" ECOG status ≤ 2
* Diagnosis of invasive or In situ breast cancer
* Patient undergoing partial mastectomy with or without axillary lymph node dissection,(without communication between the two surgical loges)

Exclusion Criteria:

* Pregnant or breast-feeding patient
* Participation at another protocol with an Investigational drug (within the last 4 weeks before enrollment)
* Known hypersensitivity to Cyanoacrylate
* Known hypersensitivity to formaldehyde
* Patient who experience systemic infections preoperatively, or have conditions that are known to interfere with the healing process
* Patient with uncontrolled diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in seroma formation | Day 3 (or 7 in case of axillary lymph node dissection), day15 and day 30 post surgery
  The volume of drain at Day 3 (or 7 in case of axillary lymph node dissection) post surgery will be documented, then patients will have an ultrasound exam at day 15 and day 30 (+or- 2 days) to measure seroma.

SECONDARY OUTCOMES:
Change in discomfort alleged by the patient | day 3 (or 7), day 15 and day 30
  Patients will be asked if they feel any discomfort in relation to seroma formation at Day 3 (or 7 in case of axillary lymph node dissection),day15 and day 30 (-or- 2 days) post surgery.

OTHER OUTCOMES:
Change in the number of needle aspiration required | day 15 and day 30
  The number of needle aspiration required at day 15 and day30 (-or- 2 days) post surgery will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Michel CONTE, MD, Principal Investigator — Hôpital Européen Marseille
Locations (2):
- France (2):
  - Centre de Chirurgie Gynecologique Et Des Maladies Du Sein, Grenoble, Auvergne-Rhône-Alpes
  - Hôpital Euroépen Marseille, Marseille, PACA